CLINICAL TRIAL: NCT07402434
Title: Advanced Diagnostic Validation and Novel Clinical Evaluation Across the CFTR Spectrum (ADVANCE-CFTR): a Prospective Study of CFTR Functional Assays, Including Rectal Organoids, to Improve the Accuracy of Diagnosing Cystic Fibrosis.
Brief Title: A Prospective Study of Advanced Diagnostics in People With an Unclear Diagnosis of Cystic Fibrosis
Acronym: ADVANCE-CFTR
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: King's College London (Other); UMC Utrecht (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 362887
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis (CF); CFTR-related Disorders
Keywords: advanced diagnostics; personalised medicine; Cystic fibrosis; CFTR-related disorders; Nasal potential difference; intestinal current measurements; organoids; sweat test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rectal biospies will be taken for both organoid formation and intestinal current measurements. Organoids will then be used for two different CFTR functional assays: Forskolin-induced swelling assays and Morphological assessment (e.g. Steady-state and high resolution 3D imaging analysis by artificial intelligence).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A - Difficult Cystic Fibrosis Diagnosis Cohort: 'Difficult-to-diagnose' patients will be recruited from the 'Difficult CF Diagnosis' service via our established referral pathway. These patients will have non-diagnostic first line CFTR testing (individuals who do not fulfil CF diagnostic criteria [2 CF-causing CFTR gene variants and/or sweat chloride concentration ≥60 mmol/L]) . These patients will be 16 years or older and will be willing to undergo a rectal biopsy.
  Interventions: Procedure: Rectal Biopsy
- Group B - Cystic Fibrosis Patient Cohort: Patients aged 16 years or older with a confirmed Cystic Fibrosis diagnosis. They would need to be willing to undergo a rectal biopsy.
  Interventions: Procedure: Rectal Biopsy
- Group C - Non-Cystic Fibrosis Patient Cohort: Patients aged 16 years or older without a Cystic Fibrosis or CFTR-related disorder diagnosis who would be willing to undergo a rectal biopsy for this study (if undergoing a lower GI endoscopy for other purposes).
  Interventions: Procedure: Rectal biopsy taken opportunistically during endoscopy procedure for other reasons.; Genetic: Blood test for CFTR Genotyping

INTERVENTIONS:
Procedure: Rectal Biopsy — Rectal biopsy sampling will be performed using either forceps or a suction device according to the method of Vonk et al (2020). Rectal biopsies will be obtained by trained and competent personnel in an appropriate setting, patients recruited will be fully informed and will have provided written consent. Once biopsy samples have been taken the resulting tissue will be processed, stored and transported using established laboratory protocols. The rectal tissue collected will be used to perform intestinal current measurements and create organoids or 'mini-organs' to allow CFTR protein function to be further characterised.
  Groups: Group A - Difficult Cystic Fibrosis Diagnosis Cohort; Group B - Cystic Fibrosis Patient Cohort
Procedure: Rectal biopsy taken opportunistically during endoscopy procedure for other reasons. — Rectal Biopsy tissue samples will be taken opportunistically for this patient cohort who are undergoing an endoscopy for other reasons. Rectal biopsies will be obtained by trained and competent personnel in an appropriate setting, patients recruited will be fully informed and will have provided written consent. The rectal tissue collected will be used to perform intestinal current measurements and create organoids or 'mini-organs' to allow CFTR protein function to be further characterised.
  Groups: Group C - Non-Cystic Fibrosis Patient Cohort
Genetic: Blood test for CFTR Genotyping — Blood test for CFTR genotyping will be taken for Group C patients to ensure these patients are 'healthy controls' and that they do not have any CFTR gene variants associated with CF.
  Groups: Group C - Non-Cystic Fibrosis Patient Cohort

SUMMARY:
Sometimes it is very difficult to tell if someone has cystic fibrosis (CF), especially when they have rare CF genes. Without this certainty, they are unlikely to get the correct treatment so their health may be affected. More accurate ways to test for CF are therefore needed in this situation. This is the aim of this study as we plan to develop a more accurate test using what are called "organoids" or "mini organs." Organoids are grown in the laboratory from a small piece of gut tissue. As they have the person's exact genes, they can show if the CF gene ("CFTR") is working correctly or not and thus if the person has CF. We will compare the organoid response with the current more established tests, such as the sweat test and CF genetics, and other recognised specialist tests called nasal potential difference (NPD) and intestinal current measurement (ICM). The gut tissue is usually taken by a quick, relatively painless, outpatient procedure (rectal biopsy). The additional benefit of organoids is that they can also help us to work out the best treatment for that individual by testing how well the gut tissue responds to different drugs in the laboratory. We wish to carry out this research to prove that gut organoids are a better way to test for CF in this situation. The goal will be to diagnose people faster and for them to get better treatment quicker, both key for leading a longer and heathier life.

DETAILED DESCRIPTION:
BACKGROUND The diagnosis of cystic fibrosis (CF) can be difficult in an important minority of individuals (~10-15% CF diagnoses), particularly when one or two rare variants of the CF gene (cystic fibrosis transmembrane conductance regulator; CFTR) are identified and the sweat test (sweat chloride concentration; SCC) is non-diagnostic. Biomarkers of CFTR function enable the quantification of individual CFTR protein function, the key underlying defect associated with CF. Such biomarkers play an important role in diagnosing CF and have the additional key capability of measuring the treatment benefits of CFTR targeting therapies, such as CFTR modulators. The currently validated biomarkers of CFTR function; such as SCC, nasal potential difference (NPD) and intestinal current measurements (ICM) can accurately characterise individuals at the extreme ranges of CFTR function (healthy and pancreatic insufficient (PI) CF), but are less reliable in intermediate ranges, particularly when clinical features are atypical. This 'difficult diagnosis' can lead to both a false positive and negative diagnostic outcome, with missed opportunities for the introduction of effective treatments, such as CFTR modulators. Some individuals remain undiagnosed for many years, even decades, so significant disease, associated with declining health, can occur. Individuals and their families are often frustrated and disillusioned by years of uncertainty. In addition, there is a group of individuals with a more limited phenotype (e.g. pancreatitis or congenital bilateral absence of the vas deferens, CBAVD), in whom the strict CF diagnostic criteria are not satisfied - their condition is termed CFTR-related disorder (RD). Recent European CF Society (ECFS) guidelines have highlighted an urgent need for a more accurate and streamlined pathway to their diagnosis.

The Difficult CF Diagnosis (DCFD) service at the Royal Brompton Hospital (RBH) uses NPD, along with whole gene analysis of CFTR and other associated genes for diagnosing unclear cases. Intestinal current measurements (ICM) - the assessment of CFTR function in Ussing chambers using ex vivo tissue biopsies of the intestinal epithelium - is currently being set-up. It is well known that an important sub-group of patients remain undiagnosed. More recently, CFTR-dependent tests in patient-derived intestinal organoids (established at the Beekman lab, University Medical Center (UMC) Utrecht University, Utrecht, The Netherlands) were also found to have excellent diagnostic capabilities with the added benefits of providing key phenotyping and prognostic information, using two different techniques - forskolin-induced-swelling (FIS) and morphological analysis (e.g. steady state lumen area, SLA). These both rely on CFTR-dependent ion and fluid secretion into the organoid lumen. Organoids can also quantify individual responses to CFTR modulators in the laboratory for estimation of potential clinical benefit and can be biobanked for future studies. How we should optimally use these different biomarkers in the context of difficult-to-diagnose individuals and treatment thereof with CFTR modulators is unclear.

ADVANCE-CFTR study is a prospective cohort study of 40-50 individuals with difficult-to-diagnose disease. They will be recruited from the Difficult CF Diagnosis (DCFD) service of the Royal Brompton Hospital. Up to 15 CF patients and 15 healthy (non-CFTR disease) controls will also be recruited to validate the tests and anchor extremes in the assays.

ELIGIBILITY:
Inclusion Criteria:

Group A: Difficult Cystic Fibrosis Diagnosis Cohort

Inclusion criteria:

1. Patients with difficult-to-diagnose CF*
2. Adults (≥16y)
3. Willing to undergo rectal biopsy
4. Able to comply with the study

   * Definition: Non-diagnostic first line CFTR testing (individuals who do not fulfil CF diagnostic criteria [2 CF-causing CFTR variants and/or sweat chloride concentration ≥60 mmol/L]). Of note, there are some individuals with <2 CF-causing CFTR variants after extended CFTR genetic analysis but with a SCC >60mmol/L. Expansion of the patient pool to include these is permissible.

Group B: Cystic Fibrosis Patient Cohort

Inclusion criteria:

1. Patients with confirmed Cystic Fibrosis
2. Adults (≥16y)
3. Willing to undergo rectal biopsy for this study
4. Able to comply with the study

Group C: Non-Cystic Fibrosis Patient Cohort

Inclusion criteria:

1. Patients without Cystic Fibrosis or CFTR-related disorder
2. Adults (≥16y)
3. Willing to undergo rectal biopsy for this study (if undergoing a lower GI endoscopy for other purposes)
4. Able to comply with the study

Exclusion Criteria:

Group A: Difficult Cystic Fibrosis Diagnosis Cohort

Exclusion criteria:

1. Contra-indication to rectal biopsy (e.g. significant bleeding diathesis)
2. History of lung transplantation
3. Receiving CFTR modulator treatment
4. Current participation (or participation within one month of enrolment) in a clinical trial of an investigational medicinal product which affects CFTR function (e.g. CFTR modulators, genetic therapies)
5. Female who is pregnant or breastfeeding
6. Unable to provide informed consent

Group B: Cystic Fibrosis Patient Cohort

Exclusion criteria:

1. Contra-indication to rectal biopsy (e.g. significant bleeding diathesis)
2. Current participation (or participation within one month of enrolment) in a clinical trial of an investigational medicinal product which affects CFTR function (e.g. CFTR modulators, genetic therapies)
3. Female who is pregnant or breastfeeding
4. Unable to provide informed consent
5. Exclude all subjects where diagnosis of CF is in doubt

Group C: Non-Cystic Fibrosis Patient Cohort

Exclusion criteria:

1. Contra-indication to rectal biopsy (e.g. significant bleeding diathesis)
2. Female who is pregnant or breastfeeding
3. Unable to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We aim to recruit 40-50 patients from the DCFD service over a 30 month period. A formal power calculation is not possible due to the exploratory nature of the analyses. Recruitment will be opportunistic, based on estimates from the DCFD service. Up to 15 healthy (non-CFTR disease) and 15 CF controls will also be recruited to validate the tests and anchor extremes in the assays.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative assessment of CFTR function | 30 months
  The primary outcome is a single or composite measurement of CFTR function derived from organoid function, Sweat Chloride Concentration (SCC), Nasal Potential Difference (NPD), and Intestinal Current Measurements (ICM). These quantitative values are then used to correlate with clinical phenotype and final diagnosis, but the outcome measure itself is CFTR functional measurement across the four test modalities.

SECONDARY OUTCOMES:
To individually phenotype patients with difficult-to-diagnose CF | 30 months
  To measure individual CFTR function in people with difficult-to-diagnose disease using multiple assays (organoids, SCC, NPD and ICM), and to correlate this with their clinical phenotype, genotype and final diagnosis.
CFTR modulator response in intestinal organoids | 30 months
  To measure CFTR modulator responses of intestinal organoids derived from individuals with difficult to-diagnose disease, taken by rectal biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Simmonds, Principal Investigator — Royal Brompton Hospital and Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilschanski M, Famini H, Strauss-Liviatan N, Rivlin J, Blau H, Bibi H, Bentur L, Yahav Y, Springer H, Kramer MR, Klar A, Ilani A, Kerem B, Kerem E. Nasal potential difference measurements in patients with atypical cystic fibrosis. Eur Respir J. 2001 Jun;17(6):1208-15. doi: 10.1183/09031936.01.00092501. PMID 11491166
- [Background] De Jonge HR, Ballmann M, Veeze H, Bronsveld I, Stanke F, Tummler B, Sinaasappel M. Ex vivo CF diagnosis by intestinal current measurements (ICM) in small aperture, circulating Ussing chambers. J Cyst Fibros. 2004 Aug;3 Suppl 2:159-63. doi: 10.1016/j.jcf.2004.05.034. PMID 15463951
- [Background] www.cftr2.com
- [Background] Waller MD, Simmonds NJ. Phenotypic variability of R117H-CFTR expression within monozygotic twins. Paediatr Respir Rev. 2016 Aug;20 Suppl:21-3. doi: 10.1016/j.prrv.2016.06.009. Epub 2016 Jun 15. PMID 27364092
- [Background] Fingeroth JM, Fossum TW. Late-onset regurgitation associated with persistent right aortic arch in two dogs. J Am Vet Med Assoc. 1987 Oct 15;191(8):981-3. PMID 3679995
- [Background] Cuyx S, Ramalho AS, Corthout N, Fieuws S, Furstova E, Arnauts K, Ferrante M, Verfaillie C, Munck S, Boon M, Proesmans M, Dupont L, De Boeck K, Vermeulen F; Belgian Organoid Project. Rectal organoid morphology analysis (ROMA) as a promising diagnostic tool in cystic fibrosis. Thorax. 2021 Nov;76(11):1146-1149. doi: 10.1136/thoraxjnl-2020-216368. Epub 2021 Apr 15. PMID 33859053
- [Background] Beekman JM, Sermet-Gaudelus I, de Boeck K, Gonska T, Derichs N, Mall MA, Mehta A, Martin U, Drumm M, Amaral MD. CFTR functional measurements in human models for diagnosis, prognosis and personalized therapy: Report on the pre-conference meeting to the 11th ECFS Basic Science Conference, Malta, 26-29 March 2014. J Cyst Fibros. 2014 Jul;13(4):363-72. doi: 10.1016/j.jcf.2014.05.007. Epub 2014 Jun 2. No abstract available. PMID 24882694
- [Background] Farrell PM, White TB, Ren CL, Hempstead SE, Accurso F, Derichs N, Howenstine M, McColley SA, Rock M, Rosenfeld M, Sermet-Gaudelus I, Southern KW, Marshall BC, Sosnay PR. Diagnosis of Cystic Fibrosis: Consensus Guidelines from the Cystic Fibrosis Foundation. J Pediatr. 2017 Feb;181S:S4-S15.e1. doi: 10.1016/j.jpeds.2016.09.064. PMID 28129811
- [Background] Hug MJ, Derichs N, Bronsveld I, Clancy JP. Measurement of ion transport function in rectal biopsies. Methods Mol Biol. 2011;741:87-107. doi: 10.1007/978-1-61779-117-8_7. PMID 21594780
- [Background] Solomon GM, Bronsveld I, Hayes K, Wilschanski M, Melotti P, Rowe SM, Sermet-Gaudelus I. Standardized Measurement of Nasal Membrane Transepithelial Potential Difference (NPD). J Vis Exp. 2018 Sep 13;(139):57006. doi: 10.3791/57006. PMID 30272672
- [Background] Dekkers JF, Alieva M, Wellens LM, Ariese HCR, Jamieson PR, Vonk AM, Amatngalim GD, Hu H, Oost KC, Snippert HJG, Beekman JM, Wehrens EJ, Visvader JE, Clevers H, Rios AC. High-resolution 3D imaging of fixed and cleared organoids. Nat Protoc. 2019 Jun;14(6):1756-1771. doi: 10.1038/s41596-019-0160-8. Epub 2019 May 3. PMID 31053799
- [Background] Vonk AM, van Mourik P, Ramalho AS, Silva IAL, Statia M, Kruisselbrink E, Suen SWF, Dekkers JF, Vleggaar FP, Houwen RHJ, Mullenders J, Boj SF, Vries R, Amaral MD, de Boeck K, van der Ent CK, Beekman JM. Protocol for Application, Standardization and Validation of the Forskolin-Induced Swelling Assay in Cystic Fibrosis Human Colon Organoids. STAR Protoc. 2020 Jun 3;1(1):100019. doi: 10.1016/j.xpro.2020.100019. eCollection 2020 Jun 19. PMID 33111074
- [Background] Rowe SM, Clancy JP, Wilschanski M. Nasal potential difference measurements to assess CFTR ion channel activity. Methods Mol Biol. 2011;741:69-86. doi: 10.1007/978-1-61779-117-8_6. PMID 21594779
- [Background] Boj SF, Vonk AM, Statia M, Su J, Vries RR, Beekman JM, Clevers H. Forskolin-induced Swelling in Intestinal Organoids: An In Vitro Assay for Assessing Drug Response in Cystic Fibrosis Patients. J Vis Exp. 2017 Feb 11;(120):55159. doi: 10.3791/55159. PMID 28287550
- [Background] Morris-Rosendahl DJ, Edwards M, McDonnell MJ, John S, Alton EWFW, Davies JC, Simmonds NJ. Whole-Gene Sequencing of CFTR Reveals a High Prevalence of the Intronic Variant c.3874-4522A>G in Cystic Fibrosis. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1438-1441. doi: 10.1164/rccm.201908-1541LE. No abstract available. PMID 32017858
- [Background] Cirilli N, Southern KW, Barben J, Vermeulen F, Munck A, Wilschanski M, Nguyen-Khoa T, Aralica M, Simmonds NJ, De Wachter E; ECFS Diagnostic Network Working Group. Standards of care guidance for sweat testing; phase two of the ECFS quality improvement programme. J Cyst Fibros. 2022 May;21(3):434-441. doi: 10.1016/j.jcf.2022.01.004. Epub 2022 Jan 19. PMID 35063396
- [Background] Dekkers JF, Berkers G, Kruisselbrink E, Vonk A, de Jonge HR, Janssens HM, Bronsveld I, van de Graaf EA, Nieuwenhuis EE, Houwen RH, Vleggaar FP, Escher JC, de Rijke YB, Majoor CJ, Heijerman HG, de Winter-de Groot KM, Clevers H, van der Ent CK, Beekman JM. Characterizing responses to CFTR-modulating drugs using rectal organoids derived from subjects with cystic fibrosis. Sci Transl Med. 2016 Jun 22;8(344):344ra84. doi: 10.1126/scitranslmed.aad8278. PMID 27334259
- [Background] de Winter-de Groot KM, Janssens HM, van Uum RT, Dekkers JF, Berkers G, Vonk A, Kruisselbrink E, Oppelaar H, Vries R, Clevers H, Houwen RHJ, Escher JC, Elias SG, de Jonge HR, de Rijke YB, Tiddens HAWM, van der Ent CK, Beekman JM. Stratifying infants with cystic fibrosis for disease severity using intestinal organoid swelling as a biomarker of CFTR function. Eur Respir J. 2018 Sep 17;52(3):1702529. doi: 10.1183/13993003.02529-2017. Print 2018 Sep. PMID 30166324
- [Background] Muilwijk D, de Poel E, van Mourik P, Suen SWF, Vonk AM, Brunsveld JE, Kruisselbrink E, Oppelaar H, Hagemeijer MC, Berkers G, de Winter-de Groot KM, Heida-Michel S, Jans SR, van Panhuis H, van der Eerden MM, van der Meer R, Roukema J, Dompeling E, Weersink EJM, Koppelman GH, Vries R, Zomer-van Ommen DD, Eijkemans MJC, van der Ent CK, Beekman JM. Forskolin-induced organoid swelling is associated with long-term cystic fibrosis disease progression. Eur Respir J. 2022 Aug 18;60(2):2100508. doi: 10.1183/13993003.00508-2021. Print 2022 Aug. PMID 35086832
- [Background] Derichs N, Sanz J, Von Kanel T, Stolpe C, Zapf A, Tummler B, Gallati S, Ballmann M. Intestinal current measurement for diagnostic classification of patients with questionable cystic fibrosis: validation and reference data. Thorax. 2010 Jul;65(7):594-9. doi: 10.1136/thx.2009.125088. PMID 20627915
- [Background] Castellani C, De Boeck K, De Wachter E, Sermet-Gaudelus I, Simmonds NJ, Southern KW; ECFS Diagnostic Network Working Group. ECFS standards of care on CFTR-related disorders: Updated diagnostic criteria. J Cyst Fibros. 2022 Nov;21(6):908-921. doi: 10.1016/j.jcf.2022.09.011. Epub 2022 Oct 8. PMID 36220763
- [Background] Simmonds NJ. Is it cystic fibrosis? The challenges of diagnosing cystic fibrosis. Paediatr Respir Rev. 2019 Aug;31:6-8. doi: 10.1016/j.prrv.2019.02.004. Epub 2019 Feb 28. PMID 30967347
- [Background] Balfour-Lynn IM, Puckey M, Simmonds NJ, Davies JC. Revisiting a diagnosis of cystic fibrosis - Uncertainties and considerations. Paediatr Respir Rev. 2022 Jun;42:29-34. doi: 10.1016/j.prrv.2021.11.002. Epub 2021 Dec 8. PMID 34998674
- [Background] Barry PJ, Simmonds NJ. Diagnosing Cystic Fibrosis in Adults. Semin Respir Crit Care Med. 2023 Apr;44(2):242-251. doi: 10.1055/s-0042-1759881. Epub 2023 Jan 9. PMID 36623819